CLINICAL TRIAL: NCT03053674
Title: Impact of Explanation Given to Parents on Rate of Post-partum Influenza Vaccination
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HYMC104-16
Record Dates: First submitted 2017-02-13; First posted 2017-02-15 (Actual); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Newborn Morbidity

STUDY DESIGN:
Intervention Model Description: Case-control study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Explanation (Experimental): Explanation to parents on importance of post-partum influenza vaccination on health of their newborn infant with a follow-up questionnaire to determine rate of vaccination
  Interventions: Other: Oral and written explanation; Other: Follow-up questionnaire
- No explanation (Active Comparator): No explanation will be given to parents but they will be followed-up with a questionnaire to determine rate of vaccination
  Interventions: Other: Follow-up questionnaire

INTERVENTIONS:
Other: Oral and written explanation — Oral and written explanation on importance of post-partum influenza vaccination for the health of their newborn infant
  Arms: Explanation
Other: Follow-up questionnaire — Follow-up questionnaire to determine whether participants have receive post-partum vaccination

SUMMARY:
The aim of this study is to determine whether an explanation to parents for the need for post-partum influenza vaccination will influence their compliance.

ELIGIBILITY:
Inclusion Criteria:

* All parents discharged from well-baby nursery

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2017-02-20 (Estimated); Primary Completion 2017-04-01 (Estimated); Study Completion 2017-07-01 (Estimated)

PRIMARY OUTCOMES:
Rate of post-partum influenza vaccination | 2 months
  Telephone questionnaire to parents to determine compliance with vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Amit Hochberg, MD, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No